CLINICAL TRIAL: NCT07308262
Title: Non-targeted Metabonomics Combined With 16S Sequencing to Analyze the Mechanism of Umbilical Moxibustion in the Treatment of IBS-B
Brief Title: Mechanism of Umbilical Moxibustion in the Treatment of IBS-b
Status: Not yet recruiting | Type: Observational
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: KY-2025-166
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Non-targeted Metabolomics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Umbilical moxibustion — Elucidate the role of the "gut microbiota-metabolite" interaction in the mechanism of umbilical moxibustion for treating IBS

SUMMARY:
Evaluate the therapeutic efficacy of umbilical moxibustion therapy for IBS. Compare and analyze the differences in gut microbiota composition and diversity between the umbilical moxibustion group and the control group based on 16S sequencing.

Compare and analyze the metabolomic differences between the umbilical moxibustion group and the control group based on non-targeted metabolomics, and identify differential metabolites associated with umbilical moxibustion treatment for IBS.

Elucidate the role of the "gut microbiota-metabolite" interaction in the mechanism of umbilical moxibustion for treating IBS.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a functional gastrointestinal disorder characterized primarily by abdominal pain and altered bowel habits. The global prevalence of IBS is approximately 11.2%, while its incidence in China ranges from 2.3% to 15.8%, with IBS-D (diarrhea-predominant IBS) being the most common subtype. This condition is characterized by recurrent episodes and is often difficult to cure. Currently, the pathogenesis of IBS remains unclear. However, as research on gut microbiota advances, increasing evidence suggests that gut microbiota plays a significant role in the development, progression, and treatment of IBS. It can contribute to the occurrence of IBS by damaging the intestinal barrier, activating immune responses, and increasing visceral sensitivity, among other mechanisms. Clinically, umbilical moxibustion therapy, which involves stimulating the Shenque point, has shown good efficacy in treating IBS, though its underlying mechanisms remain unclear. Based on non-targeted metabolomics combined with 16S rRNA gene sequencing technology, this study aims to identify biomarkers and related metabolic pathways associated with umbilical moxibustion in the treatment of IBS. The goal is to preliminarily elucidate the molecular-level mechanisms underlying the therapeutic effects of umbilical moxibustion for IBS.

ELIGIBILITY:
Study Type: Prospective, single-blinded, randomized controlled trial (patient-blinded, researcher-unblinded).

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Sample Size: 60 cases (30 in the umbilical moxibustion group, 30 in the control group), determined using G*Power (effect size d = 0.8, α = 0.05, β = 0.2; with a minimum of 26 cases per group, 15% attrition rate reserved, final 30 cases per group).
  Grouping Method: A random number table generated by SPSS 26.0 was used to allocate participants in a 1:1 ratio, with sealed envelopes employed to conceal group assignments.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Obtain the original mass spectrometry data | 12 months
  Obtain the original mass spectrometry data from metabolomics analysis, screen for differentially expressed small-molecule metabolites (meeting criteria: VIP > 1, adjusted P-value < 0.05, and fold change > 1.5), and identify no fewer than 5 potential biomarkers associated with umbilical moxibustion in the treatment of IBS-D